CLINICAL TRIAL: NCT01328184
Title: An Open-label, Two-period, Fixed-sequence Trial to Evaluate the Effect of Multiple Doses of BI 10773 on the Multiple-dose Pharmacokinetics of a Combination of Ethinylestradiol and Levonorgestrel in Healthy Premenopausal Female Volunteers
Brief Title: Drug-drug Interaction of Empagliflozin (BI 10773) and Microgynon
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1245.41; 2010-023432-16 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-04-01; First posted 2011-04-04 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
MeSH Terms: interventions — Levonorgestrel; Ethinyl Estradiol; ethinyl estradiol, levonorgestrel drug combination; empagliflozin

ARMS (2):
- Reference (Experimental): multiple doses of Microgynon
  Interventions: Drug: levonorgestrel; Drug: Ethinylestradiol
- Test (Active Comparator): multiple doses of Microgynon + BI 10773
  Interventions: Drug: levonorgestrel; Drug: Ethinylestradiol; Drug: Microgynon + BI 10773

INTERVENTIONS:
Drug: levonorgestrel — multiple doses
  Arms: Reference
Drug: levonorgestrel — multiple doses
  Arms: Test
Drug: Ethinylestradiol — multiple doses
  Arms: Test
Drug: Microgynon + BI 10773 — multiple doses BI 10773
  Arms: Test
Drug: Ethinylestradiol — multiple doses
  Arms: Reference

SUMMARY:
The objective of this study is to investigate the possible effect of multiple oral doses of 25 mg BI 10773 on the steady state pharmacokinetics of ethinylestradiol (EE) and levonogestrel (LNG) (Microgynon®).

ELIGIBILITY:
Inclusion criteria:

1. Healthy female subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1245.41.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

REFERENCES:
- [Derived] Macha S, Mattheus M, Pinnetti S, Woerle HJ, Broedl UC. Effect of empagliflozin on the steady-state pharmacokinetics of ethinylestradiol and levonorgestrel in healthy female volunteers. Clin Drug Investig. 2013 May;33(5):351-7. doi: 10.1007/s40261-013-0068-y. PMID 23512637

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Overall: A open label, two-period, fixed sequence trial. Patients received one tablet of Microgynon once daily for 14 days, immediately followed by one tablet of Microgynon once daily plus 25mg empa once daily for 7 days.
Period: Overall Study
Arm/Group | Study Overall
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Overall
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Ethinylestradiol: Area Under the Curve at Steady State Over the Uniform Dosing Interval τ (AUCτ,ss)
Description: Area under the concentration-time curve of ethinylestradiol in plasma at steady state over the uniform dosing interval τ.
Time Frame: Pre-dose, 30 min, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, and 24h after administration of Microgynon on Days 14 and 21. In addition, pre-dose samples were collected on Days 12, 13, 19, and 20.
Population: Pharmacokinetic (PK) set: Included all subjects who took at least one dose of study medication, who provided evaluable data for at least one primary PK endpoint without important protocol violations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Groups:
- Microgynon: One tablet of Microgynon once daily for 14 days.
- Microgynon Plus Empa: One tablet of Microgynon once daily plus empa 25mg once daily for seven days
Arm/Group | Microgynon | Microgynon Plus Empa
Number analyzed (Participants) | 18 | 18
pg*h/mL | 907 (24.4) | 932 (22.8)
Statistical Analysis 1: Comparison: Microgynon vs Microgynon Plus Empa; No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as Microgynon plus empa divided by Microgynon; ANOVA; Based on ANOVA with fixed term for treatment and random term for subject; Geometric Mean Ratio = 102.82, 90% CI 2-sided [97.58 to 108.35], Standard Deviation 9.0 — Standard deviation is actually the geometric coefficient of variation (gCV)

2. Primary Outcome: Levonorgestrel: Area Under the Curve at Steady State Over the Uniform Dosing Interval τ (AUCτ,ss)
Description: Area under the concentration-time curve of levonorgestrel in plasma at steady state over the uniform dosing interval τ.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Microgynon | Microgynon Plus Empa
Number analyzed (Participants) | 18 | 18
ng*h/mL | 94.0 (34.4) | 95.9 (36.6)
Statistical Analysis 1: Comparison: Microgynon vs Microgynon Plus Empa; No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as Microgynon plus empa divided by Microgynon; ANOVA; Based on ANOVA with fixed term for treatment and random term for subject; Geometric Mean Ratio = 101.94, 90% CI 2-sided [98.54 to 105.47], Standard Deviation 5.9 — Standard deviation is actually the geometric coefficient of variation (gCV)

3. Primary Outcome: Ethinylestradiol: Maximum Measured Concentration (Cmax,ss)
Description: Maximum measured concentration of ethinylestradiol in plasma at steady state over the uniform dosing interval τ.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Microgynon | Microgynon Plus Empa
Number analyzed (Participants) | 18 | 18
pg/mL | 97.6 (17.6) | 96.8 (21.8)
Statistical Analysis 1: Comparison: Microgynon vs Microgynon Plus Empa; No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as Microgynon plus empa divided by Microgynon; ANOVA; Based on ANOVA with fixed term for treatment and random term for subject; Geometric Mean Ratio = 99.22, 90% CI 2-sided [93.40 to 105.39], Standard Deviation 10.4 — Standard deviation is actually the geometric coefficient of variation (gCV)

4. Primary Outcome: Levonorgestrel: Maximum Measured Concentration (Cmax,ss)
Description: Maximum measured concentration of levonorgestrel in plasma at steady state over the uniform dosing interval τ.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Microgynon | Microgynon Plus Empa
Number analyzed (Participants) | 18 | 18
ng/mL | 7.98 (26.1) | 8.44 (25.8)
Statistical Analysis 1: Comparison: Microgynon vs Microgynon Plus Empa; No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as Microgynon plus empa divided by Microgynon; ANOVA; Based on ANOVA with fixed term for treatment and random term for subject; Geometric Mean Ratio = 105.81, 90% CI 2-sided [99.47 to 112.55], Standard Deviation 10.7 — Standard deviation is actually the geometric coefficient of variation (gCV)

5. Secondary Outcome: Ethinylestradiol: Time From Last Dosing to Maximum Measured Concentration (Tmax,ss)
Description: Time from last dosing to the maximum measured concentration of ethinylestradiol in plasma at steady state
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours(h)
Arm/Group | Microgynon | Microgynon Plus Empa
Number analyzed (Participants) | 18 | 18
hours(h) | 1.26 (39.5) [1.00 to 3.05] | 1.50 (34.2) [1.00 to 4.00]

6. Secondary Outcome: Levonorgestrel: Time From Last Dosing to Maximum Measured Concentration (Tmax,ss)
Description: Time from last dosing to the maximum measured concentration of levonorgestrel in plasma at steady state
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours(h)
Arm/Group | Microgynon | Microgynon Plus Empa
Number analyzed (Participants) | 18 | 18
hours(h) | 1.00 (28.1) [0.50 to 1.52] | 1.00 (25.5) [0.50 to 1.50]

7. Secondary Outcome: Ethinylestradiol: Apparent Clearance at Steady State (CL/Fss)
Description: Apparent clearance of ethinylestradiol in the plasma at steady state after oral administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Microgynon | Microgynon Plus Empa
Number analyzed (Participants) | 18 | 18
mL/min | 552 (24.4) | 536 (22.8)

8. Secondary Outcome: Levonorgestrel: Apparent Clearance at Steady State (CL/Fss)
Description: Apparent clearance of levonorgestrel in the plasma at steady state after oral administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Microgynon | Microgynon Plus Empa
Number analyzed (Participants) | 18 | 18
mL/min | 26.6 (34.4) | 26.1 (36.6)

9. Secondary Outcome: Ethinylestradiol: Apparent Volume of Distribution During the Terminal Phase at Steady State (Vz/Fss)
Description: Apparent volume of distribution during the terminal phase at steady state after oral administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Microgynon | Microgynon Plus Empa
Number analyzed (Participants) | 18 | 18
L | 729 (35.1) | 757 (30.3)

10. Secondary Outcome: Levonorgestrel: Apparent Volume of Distribution During the Terminal Phase at Steady State (Vz/Fss)
Description: Apparent volume of distribution during the terminal phase at steady state after oral administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Microgynon | Microgynon Plus Empa
Number analyzed (Participants) | 18 | 18
L | 84.6 (41.1) | 85.0 (38.8)

11. Secondary Outcome: Ethinylestradiol: Terminal Half-life at Steady State (t1/2,ss)
Description: Terminal half-life of ethinylestradiol in plasma at steady state
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours(h)
Arm/Group | Microgynon | Microgynon Plus Empa
Number analyzed (Participants) | 18 | 18
hours(h) | 15.3 (28.8) | 16.3 (21.8)

12. Secondary Outcome: Levonorgestrel: Terminal Half-life at Steady State (t1/2,ss)
Description: Terminal half-life of levonorgestrel in plasma at steady state
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours(h)
Arm/Group | Microgynon | Microgynon Plus Empa
Number analyzed (Participants) | 18 | 18
hours(h) | 36.7 (32.4) | 37.6 (40.7)

13. Secondary Outcome: Ethinylestradiol: Terminal Rate Constant at Steady State (λz,ss)
Description: Terminal rate constant of ethinylestradiol in plasma at steady state
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Microgynon | Microgynon Plus Empa
Number analyzed (Participants) | 18 | 18
1/h | 0.0454 (28.8) | 0.0425 (21.8)

14. Secondary Outcome: Levonorgestrel: Terminal Rate Constant at Steady State (λz,ss)
Description: Terminal rate constant of levonorgestrel in plasma at steady state
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Microgynon | Microgynon Plus Empa
Number analyzed (Participants) | 18 | 18
1/h | 0.0189 (32.4) | 0.0184 (40.7)

15. Secondary Outcome: Ethinylestradiol: Mean Residence Time at Steady State (MRTpo,ss)
Description: Mean residence time of ethinylestradiol in the body at steady state after oral administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours(h)
Arm/Group | Microgynon | Microgynon Plus Empa
Number analyzed (Participants) | 18 | 18
hours(h) | 18.6 (28.1) | 19.5 (20.5)

16. Secondary Outcome: Levonorgestrel: Mean Residence Time at Steady State (MRTpo,ss)
Description: Mean residence time of levonorgestrel in the body at steady state after oral administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours(h)
Arm/Group | Microgynon | Microgynon Plus Empa
Number analyzed (Participants) | 18 | 18
hours(h) | 48.8 (33.1) | 49.6 (41.2)

17. Secondary Outcome: Number of Participants With Clinically Relevant Abnormalities in Physical Examination, Vital Signs, ECG and Clinical Laboratory Tests.
Description: Number of participants with clinically relevant abnormalities in physical examination, vital signs and clinical laboratory tests. Relevant findings or worsenings of baseline conditions were reported as adverse events.
Time Frame: Day 1 to day 17
Population: Treated set (TS) included all subjects who took at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Microgynon | Microgynon Plus Empa
Number analyzed (Participants) | 18 | 18
participants | 0 | 0

18. Secondary Outcome: Assessment of Tolerability
Description: Tolerability will be assessed by the investigator according to the categories good, satisfactory, not satisfactory, bad and not assessable.
Time Frame: Within Day 24 to Day 31
Population: Treated set (TS) included all subjects who took at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Microgynon | Microgynon Plus Empa
Number analyzed (Participants) | 18 | 18
percentage of participants
  Good | 94.4 | 94.4
  Satisfactory | 5.6 | 5.6
  Not satisfactory | 0.0 | 0.0
  Bad | 0.0 | 0.0
  Not assessable | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: day1 to day17
Arm/Group | Microgynon | Microgynon Plus Empa
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 10/18 | 10/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Microgynon (N=18) | Microgynon Plus Empa (N=18)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 0 | 1
Thirst (General disorders) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haematoma (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes